CLINICAL TRIAL: NCT00234026
Title: Master Protocol for Mantle Cell Lymphoma A Multicenter Phase II Trial Testing Gemcitabine for the Treatment of Patients With Newly Diagnosed, Relapsed or Chemotherapy Resistant Mantle Cell Lymphoma
Brief Title: Gemcitabine in Treating Patients With Newly Diagnosed, Relapsed, or Chemotherapy-Resistant Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: SAKK 36/03; EU-20523
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Lymphoma
Keywords: recurrent mantle cell lymphoma; stage I mantle cell lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well gemcitabine works in treating patients with newly diagnosed, relapsed, or chemotherapy-resistant mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of gemcitabine, in terms of objective response and tolerability, in patients with newly diagnosed, relapsed, or chemotherapy-resistant mantle cell lymphoma.

Secondary

* Determine the time to progression and time to treatment failure in patients treated with this drug.
* Determine the response duration in patients treated with this drug.
* Determine the adverse reactions in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 3 weeks for up to 9 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually for 3 years.

PROJECTED ACCRUAL: A total of 10-29 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed mantle cell lymphoma meeting 1 of the following criteria:

  * Newly diagnosed
  * Chemotherapy resistant
  * Relapsed disease after no more than 2 prior lines of chemotherapy
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 11 mm by CT scan
* No prior or current CNS lymphoma or lymphomatous meningosis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count ≥ 1,500/mm^3 (1,000/mm^3 in case of bone marrow infiltration)
* Platelet count ≥ 100,000/mm^3 (75,000/mm^3 in case of bone marrow infiltration)

Hepatic

* Bilirubin ≤ 2 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2 times ULN
* AST and ALT ≤ 2 times ULN
* No active hepatitis

Renal

* Creatinine clearance ≥ 50 mL/min

Cardiovascular

* No congestive heart failure
* No New York Heart Association class III or IV heart disease
* No unstable angina pectoris
* No significant cardiac arrhythmia or arrhythmia requiring chronic treatment
* No myocardial infarction within the past 3 months

Immunologic

* No active autoimmune disease
* No ongoing infection (e.g., HIV)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after study participation
* No other malignancy within the past 5 years except nonmelanoma skin cancer or adequately treated carcinoma in situ of the cervix
* No uncontrolled diabetes mellitus
* No gastric ulcers
* No other uncontrolled medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent thalidomide

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Prior radiotherapy allowed provided indicator lesions were not in the irradiated field
* No concurrent radiotherapy to the lungs or mediastinum

Surgery

* Not specified

Other

* More than 30 days since prior systemic anticancer treatment
* More than 30 days since prior clinical trial participation
* No other concurrent anticancer drugs
* No other concurrent experimental drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-06; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Objective response at end of study treatment

SECONDARY OUTCOMES:
Adverse reactions at end of study treatment
Time to progression
Response duration
Time to treatment failure at end of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Felicitas Hitz, MD, Study Chair — Cantonal Hospital of St. Gallen; Lucas Widmer, MD, Principal Investigator — City Hospital Triemli
Locations (15):
- Switzerland (15):
  - Kantonspital Aarau, Aarau
  - Baden
  - Kantonsspital Baden, Baden
  - Oncology Institute of Southern Switzerland, Bellinzona
  - Spital Buelach, Bülach
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Spital Limmattal, Schlieren
  - Spital Uster, Uster
  - Kantonsspital Winterthur, Winterthur
  - Zurich
  - Onkozentrum - Klinik im Park, Zurich
  - City Hospital Triemli, Zurich
  - Klinik Hirslanden, Zurich
  - Stadtspital Waid, Zurich
  - UniversitaetsSpital Zuerich, Zurich

REFERENCES:
- [Result] Hitz F, Martinelli G, Zucca E, von Moos R, Mingrone W, Simcock M, Peterson J, Cogliatti SB, Bertoni F, Zimmermann DR, Ghielmini M; Swiss Group for Clinical Cancer Research (SAKK), Bern, Switzerland. A multicentre phase II trial of gemcitabine for the treatment of patients with newly diagnosed, relapsed or chemotherapy resistant mantle cell lymphoma: SAKK 36/03. Hematol Oncol. 2009 Sep;27(3):154-9. doi: 10.1002/hon.891. PMID 19274614